CLINICAL TRIAL: NCT01178788
Title: Progestagens for the Tertiary Prophylaxis of Preterm Delivery in Women With Short Cervix. A Randomized Multicentre Trial
Brief Title: Progestagens for the Tertiary Prophylaxis of Preterm Delivery
Acronym: PROTECT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Modena and Reggio Emilia (Other)
Responsible Party: Principal Investigator, Prof. Facchinetti Fabio, Chairman of Obstetric-Gynecology Unit, University of Modena and Reggio Emilia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2009-017441-63
Record Dates: First submitted 2010-07-08; First posted 2010-08-10 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Preterm Delivery; Neonatal Complications
Keywords: Progestagens; Tertiary Prophylaxis; Micronized Progesterone; 17 alpha hydroxy P; Preterm Delivery; Cervical shortening
MeSH Terms: conditions — Premature Birth | interventions — 17-alpha-Hydroxyprogesterone; Progesterone; Utrogestan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 17 alfa hydroxy Progesterone caproate (Active Comparator): Women treated with i.m. 17P injection/weekly (Lentogest, IBSA, Italy)
  Interventions: Drug: 17 alpha-hydroxy progesterone caproate
- Micronized Progesterone (Active Comparator): micronized P 200 mg per vagina /day (Utrogestan, Besins Healthcare, Belgium)
  Interventions: Drug: micronized Progesterone
- Control (Active Comparator): Routine clinical controls
  Interventions: Procedure: Control

INTERVENTIONS:
Drug: 17 alpha-hydroxy progesterone caproate — weekly injection of 17 P
  Other Names: Lentogest
  Arms: 17 alfa hydroxy Progesterone caproate
Drug: micronized Progesterone — daily administration of vaginal progesterone
  Other Names: Utrogestan
  Arms: Micronized Progesterone
Procedure: Control
  Other Names: Routine clinical cares
  Arms: Control

SUMMARY:
Objective: This trial would evaluate the clinical effectiveness of Progesterone(P) and 17-hydroxy Progesterone (17P) in reducing PTD, in symptomatic women at risk because of cervical shortening, in the present pregnancy.

Main outcome: Delivery before 37 weeks.

Secondary outcomes: Gestational age at delivery, Delivery <32, <35 wks, hospital admissions before delivery, birth-weight centile, NICU admission, days of NICU admission, days of oxygen supply, composite neonatal complications, congenital neonatal malformations and anomalies.

Allocated treatments will be:

Group A: 17P 341 mg i.m./weekly (Lentogest, AMSA, Italy); Group B: micronized P 200 mg per vagina /day (Utrogestan, Besins Healthcare, Belgium) Group C: no treatment, clinical observation

Concomitant treatments: Iron and folic acid supplementation, and Betamethasone (12 mg repeated once 24 hours apart) will be permitted. Is not allowed the treatment with tocolytics per os. Any treatment will be recorded.

Duration: The period of enrollment is 15 months. Cases not randomized by a clinical unit will be competitively assigned later. Results are expected 20-24 months from starting.

Sample Size: hypothesizing a risk of PTD = 0.30 efficacy is defined as a reduction to 50% (risk = 0.15). With a test potency = 0.80 and alpha = 0.025 study needs to enrol 160 patients/arm, with a total of 480 patients.

Data analysis: Methodological Unit will assign randomized treatment through a web site and it will collect data through the same way.

DETAILED DESCRIPTION:
Background: According to the last reviews Progesterone (P) and (17P) are able to reduce preterm delivery (PTD), either as prophylactic administration in the presence of previous PTD or as a treatment of the actual pregnancy, becoming at risk because of cervical shortening/preterm labour. At present is difficult to distinguish the clinical effects of P from the one of 17P as well as it is impossible to choice among the diverse doses and formulations utilized in the RCTs published so far, as well as in those under recruitment.

Protocol: Women will be treated with P, 17P or just clinically observed according to on-line randomization assignment provided by the Methodological Unit. Treatments end at the completion of 36th week. Randomization will be stratified for early (22-27+6th) and late (28-31+6th wks) PTD risk. Interim analysis will be done at 50% enrollment.

Sixty women will be allocated to each Clinical Centre to reach 480 enrollments, in the 3 arms.

Drugs will be provided by manufacturers.

ELIGIBILITY:
Inclusion Criteria:

* Women with singleton pregnancy at 22+0nd to 31+6nd week of gestation presenting with a cervical length ≤25 mm, after an episode of preterm labour.

Exclusion Criteria:

* Women with previous spontaneous PTD, multiple pregnancy, rupture of membranes, feto-maternal conditions indicating delivery, mullerian malformations, cervical surgery (cervical cerclage etc), presence of regular uterine contractions

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2010-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Preterm delivery (37 weeks of gestation) | 6 mo. after end of recruitment

SECONDARY OUTCOMES:
Delivery <32, <35 wks | 6 months after the end of the study
Hospital admissions before delivery | 6 months after the end of the study
Gestational age at delivery | 6 months after the end of the study
Birth-weight centile | 6 months after the end of the study
NICU admission | 6 months after the end of the study
days of NICU admission | 6 months after the end of the study
days of oxygen supply | 6 months after the end of the study
composite neonatal complications | 6 months after the end of the study
  Include: RDS, IVH, ROP, PVL, NEC, Sepsis
congenital neonatal anomalies | 6 months after the end of the study
congenital neonatal malformations | 6 months after the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Facchinetti, M.D., Study Chair — University of Modena and Reggio Emilia
Locations (1):
- University of Modena and Reggio Emilia, Modena, Italy

REFERENCES:
- [Derived] Facchinetti F, Vergani P, Di Tommaso M, Marozio L, Acaia B, Vicini R, Pignatti L, Locatelli A, Spitaleri M, Benedetto C, Zaina B, D'Amico R. Progestogens for Maintenance Tocolysis in Women With a Short Cervix: A Randomized Controlled Trial. Obstet Gynecol. 2017 Jul;130(1):64-70. doi: 10.1097/AOG.0000000000002065. PMID 28594783